CLINICAL TRIAL: NCT07144930
Title: Impact of Cognitive-Motor Incorporated Training and Brain Activation Patterns in Cerebrovascular Diseases With Cognitive and Motor Impairments: Post Stroke Cognitive Impairment and Moyamoya Disease
Brief Title: Cognitive-Motor Incorporated Training and Its Relations in Cerebrovascular Diseases With Cognitive and Motor Impairments
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202502047RINA
Record Dates: First submitted 2025-04-14; First posted 2025-08-28 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Moyamoya Disease; Healthy; Stroke
Keywords: Stroke; Motor-cognitive incorporated training; Cognitive function; Motor function; Post-stroke cognitive impairment
MeSH Terms: conditions — Moyamoya Disease; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- No Intervention: Healthy adults (No Intervention): Year 1: To characterize cognitive and motor performance and its relationship with brain activation patterns in individuals with post-stroke cognitive impairment (PSCI) and Moyamoya Disease (MMD).
- Individuals with post-stroke cognitive impairment (No Intervention): Year 1: To characterize cognitive and motor performance and its relationship with brain activation patterns in individuals with post-stroke cognitive impairment (PSCI) and Moyamoya Disease (MMD).
- Individuals with Moyamoya Disease (No Intervention): Year 1: To characterize cognitive and motor performance and its relationship with brain activation patterns in individuals with post-stroke cognitive impairment (PSCI) and Moyamoya Disease (MMD).
- Post-stroke cognitive impairment with MCIT program (Experimental): Year 2-3: To evaluate the short- and long-term efficacy of Motor-Cognitive Incorporated Training (MCIT) in improving cognitive and motor outcomes and modulating brain activation patterns in PSCI individuals.
  Interventions: Other: MCIT program
- Post-stroke cognitive impairment with motor training program (Active Comparator): Year 2-3: To evaluate the short- and long-term efficacy of Motor-Cognitive Incorporated Training (MCIT) in improving cognitive and motor outcomes and modulating brain activation patterns in PSCI individuals.
  Interventions: Other: Motor training program
- Moyamoya Disease with MCIT program (Experimental): Year 2-3: To evaluate the short- and long-term efficacy of MCIT in improving cognitive and motor outcomes and modulating brain activation patterns in MMD individuals.
  Interventions: Other: MCIT program
- Moyamoya Disease with motor training program (Active Comparator): Year 2-3: To evaluate the short- and long-term efficacy of MCIT in improving cognitive and motor outcomes and modulating brain activation patterns in MMD individuals.
  Interventions: Other: Motor training program

INTERVENTIONS:
Other: MCIT program — The MCIT program combines motor and cognitive training, progressing independently with increasing difficulty.
  * Motor training, based on traditional physical therapy for stroke patients, includes upper and lower extremity exercises, bed mobility, strengthening (core and extremities), and balance training, progressing from static to dynamic tasks.
  * Cognitive incorporative component, adapted from previous stroke studies, supports cognitive recovery and overall well-being. Training starts with attention and short-term memory tasks, advancing to working memory and inhibitory control with increasing difficulty. Progression requires an 80% success rate; if not achieved, tasks are simplified by reducing memory span or providing additional guidance.
  Arms: Moyamoya Disease with MCIT program; Post-stroke cognitive impairment with MCIT program
Other: Motor training program — Based on traditional physical therapy for stroke patients, includes upper and lower extremity exercises, bed mobility, strengthening (core and extremities), and balance training, progressing from static to dynamic tasks. Progression is guided by core action goals (Table 2) and depends on stable vital signs, balance, and minimal assistance. If participants are unable to progress, simpler tasks are provided.
  Arms: Moyamoya Disease with motor training program; Post-stroke cognitive impairment with motor training program

SUMMARY:
The following three-part proposal will explore the impact of applying motor-cognitive incorporated training (MCIT) in individuals with post-stroke cognitive impairment (PSCI) or Moyamoya disease (MMD), and examine the relationship between cognitive and motor impairments and brain activation patterns in these populations.

Part I is a cross-sectional study designed to characterize cognitive and motor performance and their relationship with brain activation patterns in individuals with post-stroke cognitive impairment (PSCI) or Moyamoya disease (MMD), compared to age-matched healthy controls. Thirty participants will be screened for eligibility and recruited for each group (90 participants total). After collecting basic data, all participants will undergo cognitive and motor function tests. Cognitive function tests include tests of global cognition, and executive function. Motor function tests include tests of sensorimotor function, single and dual task standing, muscle strength, and ambulation ability. Functional near-infrared spectroscopy (fNIRS) will be used to evaluate the brain activation during the cognitive tests, and single and dual task standing. Results from all tests will be used to determine the motor, cognitive, and other functional performance, and will be used in the design of the training program in Part II and III.

Part II and III are single-blinded randomized controlled trials that will explore the short and long-term effects of a motor-cognitive incorporated training (MCIT) on motor, and cognitive function in individuals with post-stroke cognitive impairment (PSCI) or Moyamoya disease (MMD). 60 individuals with PSCI (Part II), and 60 individuals with MMD (Part III) will be recruited. After screening for eligibility and collection of demographic data, participants will undergo a pretest assessment. In addition to the motor and cognitive tests used in Part I, stroke location, and time of onset will also be collected for each participant. Brain activation will be assessed during the cognitive tests, single and dual task standing assessments using fNIRS. Participants will be randomly allocated to one of the two groups (MCIT group and active control group) (n=30 in each group) via a sealed envelope selected by a blinded assistant. The training protocol is 30 minutes per session, 3 sessions per week for a total of 4 weeks. The control group will receive motor training only, including upper and lower extremity exercises, bed mobility, strengthening (core and extremities), and balance training, progressing from static to dynamic tasks. The MCIT group will engage in the program combines motor and cognitive training that starts with attention and short-term memory tasks, advancing to working memory and inhibitory control with increasing difficulty. A post-test will be conducted after the 4-week intervention, followed by follow-up assessments at 1, 3, and 12 months for individuals with PSCI or MMD in both the control group and the MCIT group. At the 3-month follow-up, participants who are unable to attend in person will be contacted by telephone. At the 12-month follow-up, all participants will receive a telephone interview focused on return-to-work status.

ELIGIBILITY:
Part 1:

Inclusion Criteria:

* For aged-matched healthy controls:

  1. being 20 years of age or older
  2. the ability to stand for more than 30 seconds
  3. a MoCA score of higher than 26.
* For PSCI participants:

  1. Diagnosis of stroke confirmed by brain CT or MRI, with symptom onset more than 7 days prior (subacute or chronic phase)
  2. Being 20 years of age or older
  3. The ability to stand for more than 30 seconds
  4. a MoCA score of less than 26
* For the MMD group:

  1. a confirmed diagnosis of Moyamoya disease or Moyamoya syndrome through CT scan or angiography
  2. If stroke occurred, being in the subacute phase (one week post-stroke)
  3. being 20 years of age or older
  4. the ability to stand for more than 30 seconds
  5. a MoCA score of less than 26

Exclusion Criteria:

1. unstable or uncontrolled vital signs, including a resting heart rate >100 or <40 BPM, a respiratory rate >20 or <12 breaths per minute, an SpO2 < 95%, a central arterial pressure (CAP) <80 mmHg, and individuals requiring ICP monitoring will also be excluded
2. requiring invasive mechanical ventilation or being deemed unsuitable by the attending physician due to unstable medical conditions
3. the presence of other neurological disorders or unstable vital signs may interfere with the experiment
4. currently hospitalized in the intensive care unit (ICU)
5. Severe visual or hearing impairments, or communication and comprehension difficulties that interfere with study participation

Part 2:

Inclusion Criteria:

1. Diagnosis of stroke confirmed by brain CT or MRI, with symptom onset more than 7 days prior (subacute or chronic phase)
2. Being 20 years of age or older
3. The ability to stand for more than 30 seconds
4. a MoCA score of less than 26

Exclusion Criteria:

1. unstable or uncontrolled vital signs, including a resting heart rate >100 or <40 BPM, a respiratory rate >20 or <12 breaths per minute, an SpO2 < 95%, a central arterial pressure (CAP) <80 mmHg, and individuals requiring ICP monitoring will also be excluded
2. requiring invasive mechanical ventilation or being deemed unsuitable by the attending physician due to unstable medical conditions
3. the presence of other neurological disorders or unstable vital signs may interfere with the experiment
4. currently hospitalized in the intensive care unit (ICU)
5. Severe visual or hearing impairments, or communication and comprehension difficulties that interfere with study participation

Part 3:

Inclusion Criteria:

1. Moyamoya disease/syndrome confirmed through CT scan or angiography
2. being in the subacute phase, defined as one week after stroke onset
3. being 20 years of age or older
4. the ability to stand for more than 30 seconds
5. a Montreal Cognitive Assessment (MoCA) score of less than 26.

Exclusion Criteria:

1. unstable or uncontrolled vital signs, including a resting heart rate >100 or <40 BPM, a respiratory rate >20 or <12 breaths per minute, an SpO2 < 95%, a central arterial pressure (CAP) <80 mmHg, and individuals requiring ICP monitoring will also be excluded
2. requiring invasive mechanical ventilation or being deemed unsuitable by the attending physician due to unstable medical conditions
3. the presence of other neurological disorders or unstable vital signs that could interfere with the experiment
4. currently hospitalized in the intensive care unit (ICU)
5. Severe visual or hearing impairments, or communication and comprehension difficulties that interfere with study participation.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Global Cognitive Function | Part 1: Baseline (Week 0); Part 2, 3: Baseline (Week 0), immediately post-intervention (Week 5), 4 weeks post-intervention (Week 9), and 12 weeks post-intervention (Week 17)
  Global cognitive function will be assessed using the Taiwan 7.1 version of the Montreal Cognitive Assessment (MoCA). The test includes 16 items and 11 categories, evaluating multiple cognitive domains. It has been validated in various clinical populations and countries. Scores range from 0 to 30, higher scores indicate better performance.
Task Switching | Part 1: Baseline (Week 0); Part 2, 3: Baseline (Week 0), immediately post-intervention (Week 5), 4 weeks post-intervention (Week 9), and 12 weeks post-intervention (Week 17)
  The Trail Making Test-A (TMT-A) requires participants to sequentially connect 25 numbered dots, while the Chinese version of TMT-B involves alternating between numbers (1-12) and Chinese zodiac signs (rat to pig). The Chinese TMT-B is a reliable tool for assessing executive function in older adults. Completion time (lower is better) is the primary outcome, with error rates also recorded.
Inhibition Control | Part 1: Baseline (Week 0); Part 2, 3: Baseline (Week 0), immediately post-intervention (Week 5), 4 weeks post-intervention (Week 9), and 12 weeks post-intervention (Week 17)
  The Chinese version of Stroop Color and Word Test (SCWT) consists of two parts: (1) a congruent condition, where participants read color-words printed in matching ink, and (2) an incongruent condition, where they identify the ink color of mismatched color-words (e.g., "black" printed in blue). Participants execute 45 seconds per task, and scores are based on the number of correct responses. Higher scores indicate better performance. The Chinese SCWT is a reliable EF assessment for older adults.
Working Memory | Part 1: Baseline (Week 0); Part 2, 3: Baseline (Week 0), immediately post-intervention (Week 5), 4 weeks post-intervention (Week 9), and 12 weeks post-intervention (Week 17)
  Digit Span Test (DS) consists of 8 items with 2 trials each, starting with 2-digit sequences and increasing to 9 digits. Participants repeat the digits in the order presented, scoring 1 point per correct response. Testing ends when both trials for an item are incorrect. Scores range from 0 to 16, with higher scores indicating better performance.
Cognitive Flexibility | Part 1: Baseline (Week 0); Part 2, 3: Baseline (Week 0), immediately post-intervention (Week 5), 4 weeks post-intervention (Week 9), and 12 weeks post-intervention (Week 17)
  Cognitive flexibility was evaluated using a Naming test. Participants name items within specific categories (fruits, vegetables, modes of transportation). They are given 1 minute to list as many items as possible from a single category, and the total number of correct responses is recorded.
Sensorimotor Function | Part 1: Baseline (Week 0); Part 2, 3: Baseline (Week 0), immediately post-intervention (Week 5), 4 weeks post-intervention (Week 9), and 12 weeks post-intervention (Week 17)
  Sensorimotor function after stroke will be measured by Fugl-Meyer Assessment for upper extremity (FMA-UE) and lower extremity (FMA-LE). The FMA-UE includes subtests evaluating the upper extremity, wrist, hand, and coordination/speed, with scores ranging from 0 to 66. The FMA-LE comprises 17 items that measure reflexes, movement, and coordination of the lower extremity, scored on a 3-point ordinal scale (0-2), with a total score of 34 points. Higher scores indicate better motor recovery. The validity and reliability of both assessments are well established.
Muscle Strength | Part 1: Baseline (Week 0); Part 2, 3: Baseline (Week 0), immediately post-intervention (Week 5), 4 weeks post-intervention (Week 9), and 12 weeks post-intervention (Week 17)
  Bilateral muscle strength of the shoulder flexors, elbow flexors, wrist extensors, ankle flexors/extensors, knee flexors/extensors, hip flexors/extensors, and hip abductors will be measured using a wireless handheld dynamometer (microFET2, Hoggan Industries, Inc., West Jordan, UT, USA). Each muscle group will be tested twice, with participants performing maximal contractions for 6 seconds per trial. A 30-second rest period will be provided between trials to prevent fatigue. The average of the two maximal efforts will be recorded.
Ambulation Ability | Part 1: Baseline (Week 0); Part 2, 3: Baseline (Week 0), immediately post-intervention (Week 5), 4 weeks post-intervention (Week 9), and 12 weeks post-intervention (Week 17)
  Ambulation ability will be evaluated using the Functional Ambulatory Category (FAC), a 6-level scale (0-5). Level 0 indicates the inability to walk, while level 5 represents complete independence. Intermediate levels reflect varying degrees of required assistance or supervision.
Dual-Task Cost (DTC) | Part 1: Baseline (Week 0); Part 2, 3: Baseline (Week 0), immediately post-intervention (Week 5), 4 weeks post-intervention (Week 9), and 12 weeks post-intervention (Week 17)
  Dual-task cost (DTC) will be calculated to perform the difference between single-task and dual-task condition, expressed as a percentage. The DTC will be calculated as: (Dual task measure - Single task measure) / Single task measure x 100%.
  For the single task, participants will stand still with a feet-together standing posture for 30 seconds, while for the dual task, they will continuously subtract 1 from a random 2-digit number while maintaining standing posture. Each condition will include a 1-minute rest period and will be repeated for three trials to ensure consistency.
  During the single and dual tasking, kinematic performance will be assessed using the 95% ellipse sway area and RMS sway, recorded by 3 wearable inertial sensors (APDM Mobility Lab® Opal system) placed bilaterally at the ankles and at the 5th lumbar vertebra. Postural sway analysis will include angle (degrees), mean velocity, acceleration, and jerk of the sway trajectory.

SECONDARY OUTCOMES:
Oxyhemoglobin [HbO] | Part 1: Baseline (Week 0); Part 2, 3: Baseline (Week 0), immediately post-intervention (Week 5), 4 weeks post-intervention (Week 9), and 12 weeks post-intervention (Week 17)
  Oxyhemoglobin [HbO] will be measured using a multichannel wearable Functional Near-Infrared Spectroscopy (fNIRS) imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NYC, USA), which emits and receives dual-wavelength near-infrared signals at 760 and 850 nm.
Deoxyhemoglobin [HbR] | Part 1: Baseline (Week 0); Part 2, 3: Baseline (Week 0), immediately post-intervention (Week 5), 4 weeks post-intervention (Week 9), and 12 weeks post-intervention (Week 17)
  Deoxyhemoglobin [HbR] will be measured using a multichannel wearable Functional Near-Infrared Spectroscopy (fNIRS) imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NYC, USA), which emits and receives dual-wavelength near-infrared signals at 760 and 850 nm.
Hemoglobin difference levels [Hbdiff] | Part 1: Baseline (Week 0); Part 2, 3: Baseline (Week 0), immediately post-intervention (Week 5), 4 weeks post-intervention (Week 9), and 12 weeks post-intervention (Week 17)
  Hemoglobin difference levels (Hbdiff) will be measured using a multichannel wearable Functional Near-Infrared Spectroscopy (fNIRS) imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NYC, USA), which emits and receives dual-wavelength near-infrared signals at 760 and 850 nm.
Activity of daily living (ADL) | Part 1: Baseline (Week 0); Part 2, 3: Baseline (Week 0), immediately post-intervention (Week 5), 4 weeks post-intervention (Week 9), and 12 weeks post-intervention (Week 17)
  The Modified Rankin Scale (mRS) assesses disability levels in ADL, ranging from 0 (no symptoms) to 6 (death). Scores between 1 and 5 reflect increasing levels of disability, from slight (independent) to severe (bedridden), with higher scores indicating lower functional ability.
Functional Independence | Part 1: Baseline (Week 0); Part 2, 3: Baseline (Week 0), immediately post-intervention (Week 5), 4 weeks post-intervention (Week 9), and 12 weeks post-intervention (Week 17)
  The Functional Independence Measure (FIM) will be used to evaluate subjects' ADL abilities. The FIM includes 18 motor and cognitive items, with total scores ranging from 18 to 126. Higher scores indicate greater independence.
Instrumental activity of daily living (IADL) | Part 1: Baseline (Week 0); Part 2, 3: Baseline (Week 0), immediately post-intervention (Week 5), 4 weeks post-intervention (Week 9), and 12 weeks post-intervention (Week 17)
  The Instrumental Activity of Daily Living (IADL) scale evaluates independence across eight domains: telephone use, shopping, food preparation, housekeeping, laundry, transportation, medication management, and financial handling. Scores range from 0 (lowest independence) to 8 (highest independence), with higher scores indicating greater functional ability.
Depression | Part 1: Baseline (Week 0); Part 2, 3: Baseline (Week 0), immediately post-intervention (Week 5), 4 weeks post-intervention (Week 9), and 12 weeks post-intervention (Week 17)
  Depression will be assessed using the Hospital Anxiety and Depression Scale (HADS), specifically the depression subscale. Scores of 8-10 indicate mild depression, 11-14 moderate, and 15-21 severe, with higher scores reflecting greater depressive symptoms.
Quality of life (QoL) | Part 1: Baseline (Week 0); Part 2, 3: Baseline (Week 0), immediately post-intervention (Week 5), 4 weeks post-intervention (Week 9), and 12 weeks post-intervention (Week 17)
  Quality of Life will be measured using the 36-item Short Form Health Survey (SF-36). The validated Taiwanese version will be used, which has strong psychometric properties. Higher scores indicate better health-related quality of life.
Return to work | Part 2, 3: 1-year post-intervention
  To track whether participants are able to return to work or re-enter their occupational environment, a telephone interview will be conducted at the 1-year follow-up. If a participant is able to return to work but requires adjustments to their job role or a change in occupation, this information will be documented in detailed notes.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Ci Liu, PhD, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University, Taipei, Taiwan